CLINICAL TRIAL: NCT00660686
Title: Exercise for Physical Health in Men With Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Lance Armstrong Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 387
Record Dates: First submitted 2008-04-11; First posted 2008-04-17 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Prostatic Neoplasm; Osteoporosis
Keywords: randomized clinical trial; elderly; cancer survivor; bone health; body composition; signs and symptoms; Androgen Deprivation Therapy
MeSH Terms: conditions — Prostatic Neoplasms; Osteoporosis; Signs and Symptoms | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Progressive resistance training program 3 times a week for 12 months
  Interventions: Behavioral: Resistance Exercise
- 2 (Active Comparator): Seated flexibility training 3 times a week for 12 months
  Interventions: Behavioral: Flexibility Training

INTERVENTIONS:
Behavioral: Resistance Exercise — 60 minute sessions 3 times a week of moderate-vigorous lower and upper body free-weight strength training plus impact training (jumps). Two of the three sessions are conducted in a supervised setting at a university fitness facility and the third session is a modified version of the exercise program performed at home. Participants are in the exercise program for 12 months
  Other Names: Arm 1: N/A
  Arms: 1
Behavioral: Flexibility Training — 60 minute session 3 times a week focusing on whole body flexibility (stretching) and relaxation (progressive neuromuscular relaxation, focused breathing) exercises. Exercises are selected to be non-weight bearing and require minimal muscle strength in order to provide a contrast to the intervention arm. Two sessions are conducted in a supervised setting at a university fitness center and the third is a home-based version of the program performed at home.
  Other Names: Arm 2: N/A
  Arms: 2

SUMMARY:
The purpose of this study is to conduct a 12-month randomized controlled trial comparing the effects of strength and impact exercise training to flexibility/relaxation training on body composition (bone, muscle and fat mass), physical function (strength, gait, power, balance and self-report physical function and symptoms) in men currently treated with hormone therapy for prostate cancer.

DETAILED DESCRIPTION:
Prostate cancer survivors with advanced disease are commonly treated with androgen deprivation therapy (ADT) to reduce testosterone. Serious side effects of ADT are rapid bone and muscle loss that can lead to osteoporosis and declines in neuromuscular function (strength, power, gait and balance) which increases the risk of fracture and falls (a risk factor for fracture) and impairs physical function. Men on ADT are 1.4 times more likely to fracture compared with their cancer-free peers and those who fracture have a poorer prognosis than those who do not. Self-report physical function is also lower among men on ADT. Exercise can prevent bone loss, neuromuscular declines and falls in several populations. However, the ability of exercise to prevent bone loss from ADT has not been tested, while data on exercise and neuromuscular function (strength only) in this population are limited to one published trial. The long-term goal of our research is to improve musculoskeletal health and function in cancer survivors. Critical first steps to meet this goal are to determine whether our previously tested program of impact and resistance exercise, shown to improve bone health and neuromuscular function in women, can prevent bone loss and neuromuscular declines in prostate cancer survivors on ADT. Based on our previous research, we have developed the Prevent Osteoporosis With Impact + Resistance (POWIR) program to be adapted to clinical populations at risk for bone loss and declines in neuromuscular function. Potentially, POWIR could mitigate bone and muscle losses from ADT, and thereby lower fracture risk and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed prostate cancer
* presently receiving or planning to begin androgen deprivation therapy for prostate cancer

Exclusion Criteria:

* Presence of bone metastases in the proximal femur and lumbar spine
* Clinically defined osteoporosis
* Current or previous use of medications known to affect bone metabolism
* Current regular participation (>2x/wk for at least 30 min/session) in a planned session of moderate-vigorous impact or resistance training
* A medical condition, disorder, or medication that contraindicates participation in moderate intensity impact or resistance exercise

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2006-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
bone mineral density, bone turnover markers (serum osteocalcin, urinary deoxypyridinoline cross-links), muscle mass, fat mass. | 12 months

SECONDARY OUTCOMES:
maximal muscle strength, gait, balance, self-report physical function, symptoms | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kerri M Winters, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU School of Nursing, Portland, Oregon, United States

REFERENCES:
- [Derived] Ernst M, Wagner C, Oeser A, Messer S, Wender A, Cryns N, Brockelmann PJ, Holtkamp U, Baumann FT, Wiskemann J, Monsef I, Scherer RW, Mishra SI, Skoetz N. Resistance training for fatigue in people with cancer. Cochrane Database Syst Rev. 2024 Nov 28;11(11):CD015518. doi: 10.1002/14651858.CD015518. PMID 39606939
- [Derived] Winters-Stone KM, Dobek JC, Bennett JA, Dieckmann NF, Maddalozzo GF, Ryan CW, Beer TM. Resistance training reduces disability in prostate cancer survivors on androgen deprivation therapy: evidence from a randomized controlled trial. Arch Phys Med Rehabil. 2015 Jan;96(1):7-14. doi: 10.1016/j.apmr.2014.08.010. Epub 2014 Sep 3. PMID 25194450